CLINICAL TRIAL: NCT03670394
Title: Capillary Refill to Detect Dehydration in Children
Brief Title: Capillary Refill for Assessment of Dehydration
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Dr. David Sheridan, Assistant professor, Oregon Health and Science University
Other Study IDs: Dehydration Assessment
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Dehydration in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Capillary Refill — We are measuring capillary refill to assess it's correlation with dehydration in children

SUMMARY:
Capillary refill is used clinically to assess multiple things in children. This is a prospective observational study of the correlation between capillary refill time and degree of dehydration in children seen in a pediatric ED.

DETAILED DESCRIPTION:
All patient presenting to the pediatric ER at OHSU less than 10 years are eligible to be enrolled if being seen for a condition putting them at risk for dehydration including emesis, diarrhea, etc. Children will have their capillary refill time measured and then sent home with a digital scale to track their weight. This will serve as the standard for calculating percent dehydration. When a patient has reached a stable weight at 1 week we will assume this is their healthy weight. There is no intervention in the study.

ELIGIBILITY:
Inclusion Criteria:

* All children with chief complaint of diarrhea, emesis, nausea, abdominal pain

Exclusion Criteria:

* Any child with chronic cardiac or pulm disease, raynauds syndrome, bilateral upper extremity trauma, previously enrolled in the study, already received IVF in the previous 48hrs, surgery within 1week, osteogenesis imperfecta.

Ages: 6 Months to 10 Years | Sex: All
Age Groups: Child
Study Population: All patients presenting to the pediatric ER at OHSu.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Capillary Refill time | 1 week
  Assessing correlation of the refill time and percent dehydration

CONTACTS AND LOCATIONS:
Overall Officials: David Sheridan, MD MR, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No